CLINICAL TRIAL: NCT06177444
Title: Post-operative Antibiotics; Effects on Risk of Infection After Cochlear Implant Surgery: A Retrospective Comparison
Brief Title: Post-operative Antibiotics; Effects on Risk of Infection After Cochlear Implant Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor
Other Study IDs: 23/46599
Record Dates: First submitted 2023-12-10; First posted 2023-12-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Infection
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative prophylactics: Patients receiving postoperative prophylactic antibiotic treatment
  Interventions: Drug: Antibiotic
- non-postoperative prophylactics: Patients NOT receiving postoperative prophylactic antibiotic treatment

INTERVENTIONS:
Drug: Antibiotic — Postoperative antibiotic treatment
  Groups: Postoperative prophylactics

SUMMARY:
Currently there is little consensus regarding postoperative antibiotic prophylactic treatment and its effect on the postoperative infection rate after Cochlear implantation. The literature on this subject is contradictory, and very limited. The aim is to assess the impact of postoperative antibiotic treatment on post-operative infection rate, and thereby discuss if postoperative antibiotic treatment has any benefits in the preventing treatment against infectious complication.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cochlear implantation at this facility from 2010 to 2022

Exclusion Criteria:

* none

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent a CI-procedure from January 2010 to December 2022, in the department of ORL at OUH, which is estimated to approximately 900 patients in total. There seems to be no study made with such a great sample-size, which therefore will have a major contribution to the knowledge on this subject.
Sampling Method: Non-Probability Sample
Enrollment: 920 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Infection rate | 1 year
  Number of infected patients

SECONDARY OUTCOMES:
Infection type | 1 year
  Number of patients with minor and severe infections

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark